CLINICAL TRIAL: NCT07133919
Title: Evaluation of the Effect of Traditional Behavior Management Techniques and AI-Assisted Child-Friendly Communication on Dental Anxiety in Pediatric Dental Anesthesia Applications
Brief Title: Effect of AI-Supported Child-Friendly Communication on Dental Anxiety in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Burak Carıkcıoglu, Associate Professor, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanakkaleOMU2
Record Dates: First submitted 2025-08-05; First posted 2025-08-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Caries, Dental; Local Anesthesia; Inferior Alveolar Nerve Block; Dental Anxiety
Keywords: dental anesthesia; dental anxiety; pediatric dentistry; pediatric patients; inferior alveolar nerve block
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Traditional Behavior Management (Control Group) (Other)
  Interventions: Behavioral: Traditional Behavior Management Techniques
- Arm 2: AI-Assisted Child-Friendly Communication (Experimental)
  Interventions: Behavioral: AI-Assisted Child-Friendly Communication

INTERVENTIONS:
Behavioral: AI-Assisted Child-Friendly Communication — AI-assisted communication tailored to the developmental stage, age, and gender of children aged 7-12 will be used. Using ChatGPT, voice recordings explaining the local anesthesia process in a child-friendly and reassuring way-avoiding anxiety-provoking terms such as "pain" and "needle"-will be prepared. Additionally, a one-minute calming and distracting story will be generated to be played during anesthesia to reduce anxiety and improve cooperation. Children will listen to the AI-generated explanation before the procedure and the story during anesthesia.
  Arms: Arm 2: AI-Assisted Child-Friendly Communication
Behavioral: Traditional Behavior Management Techniques — Before local anesthesia, traditional behavior management techniques will be applied by the pediatric dentist based on clinical experience. These include a modified Tell-Show-Do approach (avoiding direct exposure to anxiety-provoking items like dental syringes), voice control, and positive reinforcement. The anesthesia procedure will be explained verbally in an age-appropriate and reassuring manner, for example by describing the use of a "magic sleepy spray" to numb the tooth. Following this, topical anesthesia and then local anesthesia will be administered. The total procedure will not exceed 5 minutes.
  Arms: Arm 1: Traditional Behavior Management (Control Group)

SUMMARY:
This study compares the effects of traditional behavior management techniques and AI-assisted child-friendly communication on dental anxiety, physiological stress, and pain perception during local anesthesia in healthy children aged 6-12. The aim is to evaluate the effectiveness of AI-supported communication tools in reducing anxiety and improving comfort in pediatric dental treatments, potentially enhancing clinical outcomes and advancing technology use in pediatric dentistry.

DETAILED DESCRIPTION:
Successful pediatric dental treatment depends on effective therapeutic communication and tailored behavior management strategies based on the child's needs and the clinician's experience. Local anesthesia often induces dental anxiety, elevated physiological stress, and increased pain perception, which can impair treatment outcomes and contribute to dental phobia. Although traditional techniques like Tell-Show-Do and positive reinforcement are commonly used, their effectiveness may be limited in some children.

The integration of artificial intelligence (AI) and digital technologies has enabled personalized communication strategies adapted to children's cognitive and psychosocial development. AI tools such as ChatGPT act as distraction methods to reduce anxiety and stress during dental procedures. Furthermore, AI-enhanced audiovisual devices like virtual reality (VR) headsets have been shown to decrease dental anxiety, physiological stress responses, and pain perception in pediatric patients.

This study will be conducted with healthy children aged 7 to 12 who require inferior alveolar nerve block (IANB) anesthesia and have Frankl Behavior Rating Scale scores of 2 (negative) or 3 (positive). Demographic and dental data such as age, gender, and treated tooth numbers will be recorded prior to the procedure.

Participants will be randomly assigned into two groups: Group 1 (Control) and Group 2 (ChatGPT).

Control Group (Group 1):

Before local anesthesia, traditional behavior management techniques selected by the pediatric dentist based on clinical observation and experience will be applied. These include modified Tell-Show-Do (limiting exposure to potentially anxiety-provoking stimuli like dental syringes), voice control, and positive reinforcement. Explanations regarding the anesthesia procedure will be delivered verbally, tailored to the child's cognitive level and understanding capacity.

For example (From the investigators to participants):

"Hello, welcome! I see you are a bit worried, but that's very normal. People sometimes get scared of things they don't know, right? Now, please lie back comfortably, and I will tell you what are we (investigators) going to do. First, I will spray a magic sleepy water (or cold spray/warm water) on your (participants')tooth. This will make your tooth numb, so you won't feel anything. You might feel a tiny little mosquito touch, but it will pass quickly. Then your tooth will be asleep, and we (investigators) will do our work comfortably. While I'm making your tooth sleep, just lean back and think of happy memories." Following this, traditional behavior management techniques such as positive reinforcement and voice control will accompany the topical anesthesia application and then the local anesthesia procedure. The total procedure duration will not exceed 5 minutes.

Experimental Group (Group 2):

Given that cognitive abilities, language comprehension, and psychosocial needs vary by developmental stage, AI-supported communication content will be structured accordingly. Using ChatGPT, age- and gender-specific voice recordings explaining the local anesthesia procedure will be created considering developmental characteristics of children aged 7-12. Additionally, a one-minute child-friendly, anxiety-reducing story without anxiety-provoking words will be generated to be played during the anesthesia application to enhance patient cooperation and reduce anxiety.

Commands given to the AI were:

"I am about to apply local anesthesia to a [age]-year-old [girl/boy] patient with high anxiety levels. Please explain the procedure steps in a child-friendly, simple, and reassuring manner avoiding words like 'pain' and 'needle', considering developmental characteristics, age-appropriate interests, and gender-specific tendencies."

"During the anesthesia application, please tell a one-minute calming and distracting story suitable for a [age]-year-old [girl/boy], without anxiety-provoking expressions, tailored to their developmental stage and interests." Before anesthesia, children in this group will listen to the AI-generated voice explanation, and during anesthesia, the AI-generated story will be played.

Assessment criteria:

Physiological responses including heart rate and oxygen saturation will be objectively measured using a pulse oximeter (LifeNet Fingertip Pulse Oximeter; Model: KE-6004) attached to the finger before, during, and after anesthesia, recording the highest values for each phase. Subjective anxiety will be evaluated with the Venham Picture Test (VPT) and Facial Image Scale (FIS) before and after anesthesia. Pain perception will be assessed using the Wong-Baker FACES Pain Rating Scale at the end of anesthesia. Dental anxiety will be evaluated before and after anesthesia using the Modified Child Dental Anxiety Scale - Faces Version (MCDAS-f). Children's behavior during anesthesia will be recorded using the Modified Houpt Behavior Scale based on the clinician's observations. Cooperation levels will be assessed with the Frankl Behavior Rating Scale before and after anesthesia. Finally, to evaluate perceptions and attitudes toward AI-assisted communication, a 4-item child questionnaire and a 2-item parent questionnaire using 5-point Likert scales will be administered after treatment.

This study aims to compare the effectiveness of traditional behavior management techniques versus AI-assisted child-friendly communication in managing dental anxiety, physiological stress, and pain perception during local anesthesia in children, potentially contributing to innovative, evidence-based approaches in pediatric dental care.

ELIGIBILITY:
Inclusion Criteria:

* Children volunteers and their parents/legal guardians who have read and signed the informed consent form and agreed to participate in the study
* Systemically healthy children aged 6-12 years in the mixed dentition period
* Children requiring restorative dental procedures (including pulpotomy, pulp capping, or composite restorations) on mandibular teeth under inferior alveolar nerve block local anesthesia
* Children who are attending their first dental visit and demonstrate behavior rated as 2 (negative) or 3 (positive) according to the Frankl Behavior Rating Scale (Categories: 1 - definitely negative; 2 - negative; 3 - positive; 4 - definitely positive) Behaviors will be categorized as positive (+) or negative (-) based on the Frankl Behavior Rating Scale (Wright's modification)
* Children receiving local anesthesia for the first time

Exclusion Criteria:

* Children volunteers and their parents/legal guardians who read the informed consent form but declined to participate in the study
* Children with systemic diseases requiring continuous medication
* Children with mental or cognitive impairments, as well as those with visual or hearing disabilities
* Children who, after oral prophylaxis at the first visit, exhibit "definitely negative" (Frankl 1) or "definitely positive" (Frankl 4) behavior according to the Frankl Behavior Rating Scale
* Children with previous experience of local anesthesia

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pulse | 5 minutes
  Throughout the session, pulse levels were recorded using a pulse oximeter at
  three points: before, during, and after the local anesthesia.
Oxygen Saturation | 5 minutes
  Throughout the session, saturation levels were recorded using a pulse oximeter
  at three points: before, during, and after the local anesthesia.

SECONDARY OUTCOMES:
Change in Facial Image Scale (FIS)" score | Within 5 minutes before local anesthesia administration, and within 5 minutes after completion of local anesthesia procedure.
  FIS assesses anxiety in children using five facial expressions ranging from very happy to very unhappy. Children select the face that best represents their feelings at that moment. Scores range from 1 to 5; higher scores indicate higher anxiety levels.
Wong-Baker Faces Pain Rating Scale | within 5 minutes after completion of local anesthesia procedure.
  This visual self-report tool uses six faces to represent increasing levels of pain. Children choose the face that best matches their pain level. Scores range from 0 (no pain) to 10 (worst pain).
Modified Houpt Behavior Rating Scale score | During treatment
  This scale evaluates movement, crying, and overall behavior during treatment, each rated from 1 to 4. Higher total scores indicate lower cooperation and increased treatment difficulty.
Frankl Behavior Rating Scale | During treatment
  This 4-point behavioral rating scale assesses cooperation during dental treatment. Scores: 1 (definitely negative), 2 (negative), 3 (positive), 4 (definitely positive). Higher scores reflect more cooperative behavior.
Change in "Venham Picture Test (VPT)" score | Within 5 minutes before local anesthesia administration, and within 5 minutes after completion of local anesthesia procedure.
  VPT consists of 8 pairs of drawings showing children with contrasting emotional expressions. The child selects the picture they relate to most. One point is given for each anxious image selected, yielding a total score from 0 to 8; higher scores indicate more anxiety.
Change in "Modified Child Dental Anxiety Scale - faces version (MCDAS-f)" | Within 5 minutes before local anesthesia administration, and within 5 minutes after completion of local anesthesia procedure.
  MCDAS-f evaluates dental anxiety using 8 items related to specific dental procedures. Each item is rated on a 5-point Likert scale using facial images, with scores from 1 (not anxious) to 5 (very anxious). Total score ranges from 8 to 40; higher scores indicate greater anxiety.

OTHER OUTCOMES:
Perceptions and attitudes of children and parents toward AI-assisted communication | within 5 minutes after completion of local anesthesia procedure.
  This outcome measure evaluates the perceptions and attitudes of pediatric patients and their parents regarding AI-assisted communication used prior to dental treatment.
  Child questionnaire: A 4-item scale with 5-point Likert responses ("Strongly agree" to "Strongly disagree"). The items assess how the child felt after communicating with the AI before treatment, whether dental stories from the AI helped make treatment easier, whether the child would tell peers about the experience, and whether they would have allowed treatment without AI communication.
  Parent questionnaire: A 2-item scale using the same Likert format. Items assess whether AI-assisted communication helped their child cope with dental anxiety and whether they would recommend such use to others.

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Kepez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No